CLINICAL TRIAL: NCT00119236
Title: An Open-Labeled Non-Randomized Phase I Study of 17-N-allylamino-17-demethoxy Geldanamycin (17AAG) Administered With Irinotecan (CPT-11) in Patients With Advanced Solid Tumors
Brief Title: 17-AAG and Irinotecan in Treating Patients With Locally Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01467; 05-017; MSKCC-IRB-05017; NCI-7009; CDR0000434501; U01CA069856 (NIH)
Record Dates: First submitted 2005-07-12; First posted 2005-07-13 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: interventions — tanespimycin; Irinotecan

ARMS (1):
- Arm I (Experimental): Patients receive irinotecan IV over 30 minutes followed by 17-N-allylamino-17-demethoxygeldanamycin (17-AAG)* IV over 2 hours on days 1 and 8. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable or improved disease after course 2 may receive additional courses of treatment.
  Interventions: Drug: tanespimycin; Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: tanespimycin
  Other Names: 17-AAG
Drug: irinotecan hydrochloride
  Other Names: Campto; Camptosar; CPT-11; irinotecan; U-101440E

SUMMARY:
This phase I trial is studying the side effects and best dose of 17-AAG and irinotecan in treating patients with locally advanced or metastatic solid tumors. Drugs used in chemotherapy, such as 17-AAG and irinotecan, work in different ways to stop the growth of tumor cells either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (MTD) of combined 17AAG and irinotecan given weekly for two weeks in a 21-day cycle that can be used for future phase II studies.

SECONDARY OBJECTIVES:

I. To explore the effects of the combination on the expression of Hsp90 client proteins in peripheral mononuclear cells and tumor tissues. Tumor biopsies will be performed before and after 17AAG treatment in 12 patients at the MTD ("Expanded Cohort") only.

II. To investigate the clinical pharmacokinetics of intravenous 17AAG, irinotecan, and their metabolites, in this combination.

III. To obtain preliminary data on the therapeutic activity of 17AAG in combination with irinotecan in patients with advanced solid tumors.

IV. To obtain preliminary result in the relationship between tumor response and p53-status.

OUTLINE: This is an open-label, non-randomized, dose-escalation study.

Patients receive irinotecan IV over 30 minutes followed by 17-N-allylamino-17-demethoxygeldanamycin (17-AAG)* IV over 2 hours on days 1 and 8. Treatment repeats every 21 days for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients achieving stable or improved disease after course 2 may receive additional courses of treatment.

NOTE: *17-AAG is administered on days 2 and 8 during course 2 for patients treated at non-maximum tolerated doses (MTD) (dose-escalation portion) and on day 8 only during course 1 for patients treated at the MTD (expanded cohort).Cohorts of 3-6 patients receive escalating doses of 17-AAG and irinotecan until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional 12 patients are treated at the MTD.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor, excluding primary CNS tumors

  * Locally advanced or metastatic disease that is refractory to standard therapy OR for which no standard therapy exists
* Tumor assessible for biopsy by Tru-cut^®, CT guidance, or endoscopy (for patients treated at the maximum tolerated dose [expanded cohort only])

  * Pleural effusions or abdominal ascites are not considered biopsy-accessible tissue
* No known new CNS metastases that have not been previously treated
* Performance status - Karnofsky 60-100%
* WBC ≥ 3,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Bilirubin ≤ 1.5 mg/dL
* AST and ALT ≤ 3 times upper limit of normal (ULN) (5 times ULN if liver metastases are present)
* Creatinine ≤ 1.5 mg/dL
* No history of cardiac arrhythmias
* No myocardial infarction within the past 12 months
* No active ischemic heart disease within the past 12 months
* No New York Heart Association class III-IV congestive heart failure or LVEF < 40% by MUGA
* No history of uncontrolled cardiac dysrhythmia or dysrhthmias requiring medication
* No history of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation ≥ 3 beats in a row)
* No congenital long QT syndrome
* No left bundle branch block
* QTc < 450 msec (for male patients)
* QTc < 470 msec (for female patients)
* Not pregnant
* No nursing during and for 2 months after study participation
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study participation
* No serious or uncontrolled infection
* No history of serious allergic reaction to eggs or egg products
* No other medical condition that would preclude study participation
* At least 3 weeks since prior immunotherapy
* No concurrent prophylactic filgrastim (G-CSF) or sargramostim (GM-CSF)
* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin)
* Prior irinotecan allowed
* No prior 17-N-allylamino-17-demethoxygeldanamycin (17-AAG)
* At least 2 weeks since prior non-myelosuppressive chemotherapy (at the discretion of the principal investigator)
* At least 3 weeks since prior radiotherapy
* No prior radiotherapy field that included the heart (e.g., mantle)
* Recovered from all prior therapy
* At least 3 weeks since prior anticancer investigational therapeutic drugs
* More than 7 days since prior and no concurrent inducers, inhibitors, or modifiers of CYP3A4, including any of the following:

  * Fluconazole
  * Itraconazole
  * Ketoconazole
  * Azithromycin
  * Clarithromycin
  * Erythromycin
  * Troleandomycin
  * Nifedipine
  * Verapamil
  * Diltiazem
  * Nefazodone
  * Cyclosporine
  * Grapefruit juice (> 1 quart/day)
  * Indinavir
  * Nelfinavir
  * Ritonavir
  * Saquinavir
  * Carbamazepine
  * Phenobarbital
  * Phenytoin
  * Rifampin
  * Hydrastis canadensis (goldenseal)
  * Hypericum perforatum (St. John's wort)
  * Uncaria tomentosa (cat's claw)
  * Echinacea angustifolia root
  * Trifolium pratense (wild cherry)
  * Matricaria chamomila (chamomile)
  * Glycyrrhiza glabra (licorice)
  * Dillapiol
  * Hypericin
  * Naringenin
* No concurrent medications that would prolong QTc
* No concurrent vitamins, antioxidants, herbal preparations, or supplements

  * Concurrent single daily multivitamin allowed
* No other concurrent anticancer therapy
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2005-05; Primary Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determined by dose-limiting toxicities | 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Archie Tse, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States